CLINICAL TRIAL: NCT01754935
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of VX-509 Using Magnetic Resonance Imaging and Arthroscopic Biopsies in Subjects With Active Rheumatoid Arthritis on Stable Disease-Modifying Antirheumatic Drugs
Brief Title: A Magnetic Resonance Imaging Study and Arthroscopic Biopsy Substudy in Subjects With Active Rheumatoid Arthritis Receiving VX-509, an Oral JAK3 Inhibitor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX12-509-103; 2012-003439-41 (EudraCT Number)
Record Dates: First submitted 2012-12-18; First posted 2012-12-21 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — 2-((2-(1H-pyrrolo(2,3-b)pyridin-3-yl)pyrimidin-4-yl)amino)-2-methyl-N-(2,2,2-trifluoroethyl)butanamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- VX-509 100 mg qd Arm (Experimental)
  Interventions: Drug: VX-509
- VX-509 200 mg qd Arm (Experimental)
  Interventions: Drug: VX-509
- VX-509 300 mg qd Arm (Experimental)
  Interventions: Drug: VX-509
- Placebo Arm (Placebo Comparator)
  Interventions: Drug: VX-509 matching placebo

INTERVENTIONS:
Drug: VX-509 — 50 mg oral tablet
  Arms: VX-509 100 mg qd Arm; VX-509 200 mg qd Arm; VX-509 300 mg qd Arm
Drug: VX-509 matching placebo — 0 mg oral tablet
  Arms: Placebo Arm

SUMMARY:
The current study is designed to evaluate the safety and efficacy, including MRI imaging, across a range of VX-509 doses in subjects with active rheumatoid arthritis (RA) who have had an inadequate response to disease-modifying antirheumatic drugs (DMARDs).

DETAILED DESCRIPTION:
VX-509 is an oral, selective Janus kinase 3 (JAK3) inhibitor being developed by Vertex. In autoimmune diseases, JAK3 is an essential component of the immune signaling cascade. This cascade ultimately contributes to abnormal immune response that results in chronic inflammation and, in the case of rheumatoid arthritis (RA), irreversible damage to cartilage and bones. Selective inhibition of JAK3 offers a new disease modifying approach to the treatment of RA, and a broad range of other autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 to 65 years of age (inclusive)
* Diagnosis of RA
* Swollen joint count of ≥6 out of 66 joints and tender joint count of ≥6 out of 68 joints
* Seropositivity based on either a positive rheumatoid factor or anti cyclic citrullinated peptide antibody at screening -OR- known erosive disease based on previous X-ray report or erosions detected on screening hand and foot X-ray
* Baseline CRP level or Westergren erythrocyte sedimentation rate ≥1.2 × upper limit of normal
* Receiving stable therapy with 1 of the following DMARDs: methotrexate, sulfasalazine, leflunomide, anti-malarial drug, or penicillamine
* Palpable 2+ synovitis of the wrist or ≥2 MCPs in the MRI-designated hand

Exclusion Criteria:

* History or presence of a clinically significant medical disorder other than RA that, in the opinion of the investigator and medical monitor, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.
* Inflammatory, rheumatological disorders other than RA, where arthritis may be a prominent feature
* Planned surgery during the study
* History of alcohol or drug abuse, or excessive alcohol consumption
* History of tuberculosis (TB) infection of any kind (pulmonary or extrapulmonary, active or latent), regardless of history of anti-TB treatment.
* Pregnant or nursing an infant or with a life partner who is pregnant, nursing, or planning to become pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving a ≥20% improvement in disease severity according to the American College of Rheumatology criteria (ACR20), using C reactive protein (CRP) (ACR20 CRP) | Week 12
Change from baseline in Disease Activity Score 28 using CRP (4-component) (DAS28-4[CRP]) | Week 12
Change from baseline in OMERACT RAMRIS synovitis score in designated hand wrist | Week 12
Change from baseline in OMERACT RAMRIS bone marrow edema (osteitis) in designated hand wrist | Week 12
Change from baseline in OMERACT RAMRIS erosion score in designated hand wrist | Week 12

SECONDARY OUTCOMES:
Proportion of subjects achieving a ACR50 CRP and ACR70 CRP responses | Week 12
Proportion of subjects with DAS28 CRP <2.6, and those who achieve a remission, moderate response or good response according to the European League Against Rheumatism (EULAR) response criteria | Week 12
ACR hybrid scores | Week 12
Change from baseline in Health Assessment Questionnaire -Disability Index (HAQ-DI) | Week 12
Change from baseline in OMERACT RAMRIS synovitis, bone marrow edema (osteitis), erosion scores | Week 6
PK parameters of VX-509 and its metabolite in plasma (maximum observed concentration [Cmax] and area under the concentration versus time curve [AUC]) | Week 12
Safety and tolerability as indicated by adverse events, laboratory tests, electrocardiograms (ECGs) and vital signs | Week 12
Change from baseline in the Physical Function subscale of the 36-item Short Form (SF-36) | Week 12
Change from baseline in the Physical Component and Mental Health Components of the SF-36 | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Bloom, MD, FACR, FAAP, Study Chair — Vertex Pharmaceuticals Incorporated
Locations (30):
- United States (21):
  - Vertex Investigational Site, Stanford, California
  - Vertex Investigational Site, Upland, California
  - Vertex Investigational Site, Fort Lauderdale, Florida
  - Vertex Investigational Site, Venice, Florida
  - Vertex Investigational Site, West Palm Beach, Florida
  - Vertex Investigational Site, Canton, Georgia
  - Vertex Investigational Site, Decatur, Georgia
  - Vertex Investigational Site, Kansas City, Kansas
  - Vertex Investigational Site, Elizabethtown, Kentucky
  - Vertex Investigational Site, Frederick, Maryland
  - Vertex Investigational Site, Lincoln, Nebraska
  - Vertex Investigational Site, Rochester, New York
  - Vertex Investigational Site, Greenboro, North Carolina
  - Vertex Investigational Site, Duncansville, Pennsylvania
  - Vertex Investigational Site, Charleston, South Carolina
  - Vertex Investigational Site, Memphis, Tennessee
  - Vertex Investigational Site, Katy, Texas
  - Vertex Investigational Site, San Antonio, Texas
  - Vertex Investigational Site, Webster, Texas
  - Vertex Investigational Site, Seattle, Washington
  - Vertex Investigational Site, Spokane, Washington
- Denmark (2):
  - Vertex Investigational Site, Hillerød
  - Vertex Investigational Site, Hjørring
- Vertex Investigational Site, Tallinn, Estonia
- Vertex Investigational Site, Vilnius, Lithuania
- Netherlands (2):
  - Vertex Investigational Site, Heerlen
  - Vertex Investigational Site, Utrecht
- South Africa (3):
  - Vertex Investigational Site, Johannesburg
  - Vertex Investigational Site, Pretoria
  - Vertex Investigational Site, Stellenbosch

REFERENCES:
- [Derived] Genovese MC, Yang F, Ostergaard M, Kinnman N. Efficacy of VX-509 (decernotinib) in combination with a disease-modifying antirheumatic drug in patients with rheumatoid arthritis: clinical and MRI findings. Ann Rheum Dis. 2016 Nov;75(11):1979-1983. doi: 10.1136/annrheumdis-2015-208901. Epub 2016 Apr 15. PMID 27084959